CLINICAL TRIAL: NCT02850835
Title: Role of Video Decision Aid in Pelvic Organ Prolapse Treatment Selection in Latina Women
Brief Title: Video Decision Aid in Latina Women With Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Teodoro Ignacio Montoya, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E16059
Record Dates: First submitted 2016-07-07; First posted 2016-08-01 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Decision Aid; Pelvic Organ Prolapse (POP)
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Decision Aid (Experimental): This group will be shown a video decision aid along with their standard of care.
  Interventions: Other: Video Decision Aid
- Standard Care (No Intervention): This group will not see the video decision aid and will only receive standard of care.

INTERVENTIONS:
Other: Video Decision Aid — A video decision aid was developed inform patients about pelvic organ prolapse, to include female anatomy, and treatment options.
  Other Names: VDA
  Arms: Video Decision Aid

SUMMARY:
Pelvic organ prolapse (POP) is a highly prevalent condition among women that impairs quality of life, daily activities and sexual function. Latina women are disproportionally affected, with significantly higher rates of POP compared to women of other ethnicities. Decision aids have been used to increase patient knowledge prior to physician intervention and to facilitate informed patient participation on treatment selection. The investigators hypothesize that the use of a video decision aid prior to initial Urogynecology specialist evaluation of Latina women with POP in a border region university-affiliated medical clinic, will increase patient knowledge regarding the condition, decrease decisional conflict regarding selection among different treatment options and increase patient satisfaction with selected treatment.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a highly prevalent condition among women that impairs quality of life, daily activities and sexual function. Latina women are disproportionally affected, with significantly higher rates of POP compared to women of other ethnicities. Counseling Latina women suffering from POP is often complex due to a variety of factors, including language barriers, limited patient understanding of anatomy and disease etiology and confusion regarding surgical versus nonsurgical treatment options. Decision aids have been used to increase patient knowledge prior to physician intervention and to facilitate informed patient participation on treatment selection. The investigators hypothesize that the use of a video decision aid prior to initial Urogynecology specialist evaluation of Latina women with POP will increase patient knowledge regarding the condition, decrease decisional conflict regarding selection among different treatment options and increase patient satisfaction with selected treatment, empowering these women as active participants in their healthcare instead of relying on provider input alone.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic Women
* Referred for evaluation of pelvic organ prolapse for the first time

Exclusion Criteria:

* Women previously referred or treated for pelvic organ prolapse
* Women who do not live in El Paso, Texas

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline decisional conflict score at 6 months. | 6 months
  Decisional Conflict Scale will be used

SECONDARY OUTCOMES:
Change from baseline knowledge of condition score at 6 months. | 6 months
  12-item questionnaire of female pelvic anatomy and pelvic organ prolapse concepts will be used
Change from baseline satisfaction with selected treatment at 6 months. | 6 months
  Satisfaction with Decision Scale-(PFD) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Teodoro I Montoya, M.D., Principal Investigator — Texas Tech University Health Sciences Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Buchsbaum GM, Duecy EE, Kerr LA, Huang LS, Perevich M, Guzick DS. Pelvic organ prolapse in nulliparous women and their parous sisters. Obstet Gynecol. 2006 Dec;108(6):1388-93. doi: 10.1097/01.AOG.0000245784.31082.ed. PMID 17138771
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Jelovsek JE, Barber MD. Women seeking treatment for advanced pelvic organ prolapse have decreased body image and quality of life. Am J Obstet Gynecol. 2006 May;194(5):1455-61. doi: 10.1016/j.ajog.2006.01.060. PMID 16647928
- [Background] Andersen R, Lewis SZ, Giachello AL, Aday LA, Chiu G. Access to medical care among the Hispanic population of the southwestern United States. J Health Soc Behav. 1981 Mar;22(1):78-89. No abstract available. PMID 7240708
- [Background] Herman JP, Blangero A, Madelain L, Khan A, Harwood MR. Saccade adaptation as a model of flexible and general motor learning. Exp Eye Res. 2013 Sep;114:6-15. doi: 10.1016/j.exer.2013.04.001. Epub 2013 Apr 15. PMID 23597598
- [Background] O'Connor AM, Rostom A, Fiset V, Tetroe J, Entwistle V, Llewellyn-Thomas H, Holmes-Rovner M, Barry M, Jones J. Decision aids for patients facing health treatment or screening decisions: systematic review. BMJ. 1999 Sep 18;319(7212):731-4. doi: 10.1136/bmj.319.7212.731. PMID 10487995
- [Derived] Montoya TI, Rondeau NU, Maldonado PA, Mallett VT. Decision Aid Video for Treatment Selection in Latinas With Symptomatic Pelvic Organ Prolapse: A Randomized Pilot Study. Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):39-45. doi: 10.1097/SPV.0000000000000727. PMID 31008776